CLINICAL TRIAL: NCT01156116
Title: Effective Treatment of Sleep Apnea in Prediabetes to Reduce Cardiometabolic Risk
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 09-249-A
Record Dates: First submitted 2010-06-23; First posted 2010-07-02 (Estimated); Results first posted 2015-05-27 (Estimated); Last update posted 2015-05-27 (Estimated); Status verified 2015-05

CONDITIONS: Diabetes; Sleep Apnea
Keywords: CPAP; diabetes; sleep apnea
MeSH Terms: conditions — Diabetes Mellitus; Sleep Apnea Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Continuous positive airway pressure (Active Comparator): 2 weeks of continuous positive airway pressure (CPAP) treatment which includes wearing the CPAP mask for 8 hours each night
  Interventions: Device: CPAP mask
- Placebo (Placebo Comparator): 2 weeks of oral administration of a placebo tablet 30min before bedtime
  Interventions: Drug: Placebo

INTERVENTIONS:
Device: CPAP mask — The subjects who are randomized to CPAP treatment will undergo an overnight CPAP titration in the laboratory, which will be performed manually by a registered technician according to American Academy of Sleep Medicine (AASM) guidelines .Subjects will be admitted in the early evening and will receive positive airway pressure education, hands on demonstration, careful mask fitting and acclimatization prior to titration. The goal during the titration will be to determine the optimal CPAP pressure setting that eliminates obstructive respiratory events, restore oxygen saturations and sleep continuity.
  ________________________________________
  Other Names: continuous positive airway pressure therapy
  Arms: Continuous positive airway pressure
Drug: Placebo — oral placebo tablet
  Arms: Placebo

SUMMARY:
Although obstructive sleep apnea (OSA) is associated with impaired glucose tolerance and diabetes, it remains unclear whether OSA treatment with continuous positive airway pressure (CPAP) has metabolic benefits. The objective of this study is to determine the effect of 8-hour nightly CPAP treatment on glucose metabolism in individuals with prediabetes and OSA.

DETAILED DESCRIPTION:
Although obstructive sleep apnea (OSA) is associated with impaired glucose tolerance and diabetes, it remains unclear whether OSA treatment with continuous positive airway pressure (CPAP) has metabolic benefits. To determine the effect of 8-hour nightly CPAP treatment on glucose metabolism in individuals with prediabetes and OSA. In a randomized, controlled parallel group study, 39 participants were randomized (2:1) to receive either 8-hour nightly CPAP (n=26) or oral placebo (n=13). Sleep was polysomnographically recorded in the laboratory on each night. CPAP adherence was ensured by continuous supervision. Participants continued their daily daytime routine activities outside the laboratory. Glucose metabolism was assessed at baseline and after 2-weeks of assigned treatment using both the oral and intravenous glucose tolerance tests (OGTT and ivGTT, respectively). The primary outcome was the overall glucose response as quantified by the area under the curve for glucose during 2-hour oral glucose tolerance testing.

ELIGIBILITY:
Inclusion Criteria:

* Overweight or obese adults (age ≥45 yrs and BMI ≥25 kg/m2)
* prediabetes and OSA (AHI ≥ 5)
* regular life styles and schedules (no shift work in the past 6 months, no travel across time zones during the past 4 weeks)
* habitual bedtimes of at least 6 hours but not exceeding 9 hours will be eligible.
* not to take any medications during the study period with the exception of antihypertensives and lipid lowering agents
* not on hormone replacement therapy.
* have sedentary activities and no competitive athletes or subjects with high exercise levels.

Exclusion Criteria:

* previous or current treatment with supplemental oxygen
* requirement of supplemental oxygen or bi-level positive airway pressure for OSA treatment during titration
* presence of active infection, psychiatric disease or history of other significant illness (e.g., myocardial infarction, congestive heart failure, stroke, arrhythmia, chronic kidney or liver disease0
* clinical depression as evidenced by a score >16 in CES-D scale
* smoking, or routine alcohol use (more than 2 drinks per day), or excessive caffeine intake (>300mg per day)

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2009-10; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Esra Tasali, MD, Principal Investigator — University of Chicago
Locations (1):
- The University of Chicago, Chicago, Illinois, United States

REFERENCES:
- [Derived] Pamidi S, Chapotot F, Wroblewski K, Whitmore H, Polonsky T, Tasali E. Optimal Continuous Positive Airway Pressure Treatment of Obstructive Sleep Apnea Reduces Daytime Resting Heart Rate in Prediabetes: A Randomized Controlled Study. J Am Heart Assoc. 2020 Oct 20;9(19):e016871. doi: 10.1161/JAHA.120.016871. Epub 2020 Oct 1. PMID 32998624
- [Derived] Pamidi S, Wroblewski K, Stepien M, Sharif-Sidi K, Kilkus J, Whitmore H, Tasali E. Eight Hours of Nightly Continuous Positive Airway Pressure Treatment of Obstructive Sleep Apnea Improves Glucose Metabolism in Patients with Prediabetes. A Randomized Controlled Trial. Am J Respir Crit Care Med. 2015 Jul 1;192(1):96-105. doi: 10.1164/rccm.201408-1564OC. PMID 25897569

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Continuous Positive Airway Pressure | Placebo
Started | 26 | 13
Completed | 21 | 12
Not Completed | 5 | 1
Not completed — Withdrawal by Subject | 3 | 1
Not completed — CPAP intolerance | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Continuous Positive Airway Pressure | Placebo | Total
Number analyzed (Participants) | 26 | 13 | 39
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.8 (6.2) | 55.2 (8.4) | 54.3 (6.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 3 | 13
  Male | 16 | 10 | 26
Region of Enrollment [Number; unit: participants]
  United States | 26 | 13 | 39

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Area Under the Curve (AUC) Glucose at Week 2
Description: The area under the glucose time curve, between 0 and 120 minutes of the OGTT, was calculated for each patient using the trapezoidal rule .
  Change = Week 2 - Baseline.
Time Frame: Baseline and Week 2
Population: One patient in the Placebo group who withdrew prior to any testing was excluded from the analysis.
Measure: Mean (95% Confidence Interval); unit: (mg/dL)*min
Arm/Group | Continuous Positive Airway Pressure | Placebo
Number analyzed (Participants) | 26 | 12
(mg/dL)*min | -794.2 [-1446.4 to -142.0] | 482.7 [-422.2 to 1387.7]
Statistical Analysis 1: Comparison: Continuous Positive Airway Pressure vs Placebo; Test type: Superiority or Other; p = 0.03, Mixed Models Analysis; Analyses were adjusted for age, body mass index, and ethnicity-based diabetes risk

2. Secondary Outcome: Change From Baseline in Insulin Sensitivity (SI) at Week 2
Description: SI is estimated from modeling of the insulin and glucose values during the intravenous glucose tolerance test (ivGTT).
  Change = Week 2 - Baseline.
Time Frame: Baseline and Week 2
Population: One patient from each group was excluded from the analysis since they were missing SI data at both Baseline and Week 2.
Measure: Mean (95% Confidence Interval); unit: [mU/L]^-1·[min]^-1
Arm/Group | Continuous Positive Airway Pressure | Placebo
Number analyzed (Participants) | 25 | 12
[mU/L]^-1·[min]^-1 | 0.31 [-0.11 to 0.74] | -0.46 [-1.07 to 0.15]
Statistical Analysis 1: Comparison: Continuous Positive Airway Pressure vs Placebo; Test type: Superiority or Other; p = 0.04, Mixed Models Analysis; Analyses were adjusted for age, body mass index, and ethnicity-based diabetes risk

3. Secondary Outcome: Change From Baseline in 24-hr Systolic Blood Pressure (mmHg) at Week 2
Description: The average systolic blood pressure measured over a 24-hr period was calculated for each patient.
  Change = Week 2 - Baseline.
Time Frame: Baseline and Week 2
Population: Patients were excluded from the analysis if they were missing blood pressure data at both Baseline and Week 2.
Measure: Mean (95% Confidence Interval); unit: mmHg
Arm/Group | Continuous Positive Airway Pressure | Placebo
Number analyzed (Participants) | 22 | 10
mmHg | -1.9 [-6.2 to 2.3] | 7.6 [1.9 to 13.3]
Statistical Analysis 1: Comparison: Continuous Positive Airway Pressure vs Placebo; Test type: Superiority or Other; p = 0.009, Mixed Models Analysis; Analyses were adjusted for age, body mass index, and ethnicity-based diabetes risk

4. Secondary Outcome: Change From Baseline in 24-hr Diastolic Blood Pressure (mmHg) at Week 2
Description: The average diastolic blood pressure over a 24-hr period was calculated for each patient.
  Change = Week 2 - Baseline
Time Frame: Baseline and Week 2
Population: Patients were excluded from the analysis if they were missing blood pressure data at both Baseline and Week 2.
Measure: Mean (95% Confidence Interval); unit: mmHg
Arm/Group | Continuous Positive Airway Pressure | Placebo
Number analyzed (Participants) | 22 | 10
mmHg | -2.6 [-4.9 to -0.3] | 4.5 [1.4 to 7.5]
Statistical Analysis 1: Comparison: Continuous Positive Airway Pressure vs Placebo; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; Analyses were adjusted for age, body mass index, and ethnicity-based diabetes risk

ADVERSE EVENTS:
Time Frame: 2 weeks
Description: Only treatment related adverse events were collected.
Arm/Group | Continuous Positive Airway Pressure | Placebo
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/13
Other Adverse Events (participants affected / at risk) | 0/26 | 0/13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes